CLINICAL TRIAL: NCT05413746
Title: Proof of Concept: Prospective Study of the New REOXCARE Dressing to Improve Healing in Diabetic Foot Ulcers (DFU)
Brief Title: REOXCARE Dressing to Improve Healing in Diabetic Foot Ulcers (DFU)
Acronym: REOXDFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Histocell, S.L. (Industry)
Collaborators: Hospital de Cruces (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REOXCARE.DFU
Record Dates: First submitted 2022-06-01; First posted 2022-06-10 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus; Foot Ulcer; Neuroischemic Foot Ulcer
Keywords: Wound care; Diabetic foot ulcer; Antioxidants
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antioxidant dressing (active product) (Experimental): Wound bed debridement, Antioxidant dressing (active product) application in the wound bed, covered with secondary dressing.
  Device: Reoxcare®
  Interventions: Device: Reoxcare antioxidant dressing

INTERVENTIONS:
Device: Reoxcare antioxidant dressing — After wound cleaning activities, wound bed debridement if necessary and elimination of hyperkeratotic edges, wounds are treated with Reoxcare as primary dressing and the approppriate secondary dressing for adequate exudates management

SUMMARY:
It has been shown that diabetic patients present a significant increase in markers related to oxidative stress, which increases even more in those with diabetic foot ulcers and gradually depending on the severity of the injury and inversely to the mechanisms of physiological antioxidants of these patients. Therefore, these patients present a situation of oxidative stress (high lipid peroxidation), with an insufficient level of antioxidant enzymes to reverse this state, which leads to maintenance of the inflammatory situation and therefore the chronification of the ulcer. Investigators' aim in this study is to measure the benefits that the application of the product with antioxidant capacity REOXCARE can bring, together with the usual good clinical wound care guidelines and other essential therapeutic activities, such as pressure relief in the area of the ulcers.

DETAILED DESCRIPTION:
The frequency in the appearance of diabetic foot lesions is extremely high; it is estimated that around 15% of people with diabetes will present some compromise at the level of the foot during the evolution of the disease. The high rate of recurrence of these lesions and their high mortality rate make this pathology an important health problem with high health, economic and social repercussions. Diabetic foot injury is defined as any infection, ulceration, and/or destruction of the deep tissues of the foot associated with neurological, vascular, and metabolic disorders (sustained hyperglycemia) in the lower limbs of people with diabetes. Between 40% and 70% of lower-limb amputations occur in the diabetic population, and in up to 85% of cases, the triggering factor is ulcer, associated with infection and gangrene. The incidence of a new episode after an amputation is around 50% 5 years later.

It has been shown that diabetic patients present a significant increase in markers related to oxidative stress, which increases even more in those with diabetic foot ulcers and gradually depending on the severity of the injury and inversely to the mechanisms of physiological antioxidants of these patients. Therefore, these patients present a situation of oxidative stress (high lipid peroxidation), with an insufficient level of antioxidant enzymes to reverse this state, which leads to maintenance of the inflammatory situation and therefore the chronification of the ulcer. Investigators' aim in this study is to measure the benefits that the application of the product with antioxidant capacity REOXCARE can bring, together with the usual good clinical wound care guidelines and other essential therapeutic activities, such as pressure relief in the area of the ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Post-surgical diabetic foot ulcers after an amputation process, with the purpose of closure by "secondary intention". There may be prior limb bypass surgery.
* Diabetic foot ulcers with a neuroischemic component
* Ulcers located on the foot, below the malleoli.
* Ulcers without clinical signs of infection at the time of recruitment
* Patients with sufficient physical and health characteristics to be able to respond to treatment and over 18 years of age.
* The patient and/or his/her relative/representative have given their informed consent in writing.
* In the case of several lesions in the same patient that meet the inclusion criteria, select, at the investigator's discretion, the ulcer that can best benefit from the treatment. The rest of the injuries will be treated according to clinical criteria, with the dressings available in the usual clinical practice of the Center or REOXCARE.

Exclusion Criteria:

* Patients with wounds with clinical signs of local infection
* Intolerance to the components of the product under study.
* Uncontrolled diabetes
* Other ulcers not included in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Changes in Granulation tissue in the wound bed | At baseline, after 1 week, after 2 week, after 3 week, after 4 weeks, after 5 weeks, after 6 weeks, after 7 weeks and after 8 week
  The percentage of granulation tissue in the wound bed is estimated by the clinicians in each week of Reoxcare treatment, At baseline and every week
Changes in wound size | At baseline, after 1 week, after 2 week, after 3 week, after 4 weeks, after 5 weeks, after 6 weeks, after 7 weeks and after 8 week
  The difference in wound area between first and last dressing Reoxcare treatment

SECONDARY OUTCOMES:
Number of completely healed wounds | At baseline, after 1 week, after 2 week, after 3 week, after 4 weeks, after 5 weeks, after 6 weeks, after 7 weeks and after 8 week
  Number of wounds closed with respect to total number of wounds at each frame time
Time to removal of non-viable tissue from wound bed | At baseline, after 1 week, after 2 week, after 3 week, after 4 weeks, after 5 weeks, after 6 weeks, after 7 weeks and after 8 week
  Percentage of wounds with non-viable tissue in the wound bed at each frame time

CONTACTS AND LOCATIONS:
Overall Officials: Andima Basterretxea, MD, Principal Investigator — Hospital Universitario de Cruces
Locations (2):
- Spain (2):
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Histocell, Derio, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro B, Palomares T, Azcoitia I, Bastida F, del Olmo M, Soldevilla JJ, Alonso-Varona A. Development and preclinical evaluation of a new galactomannan-based dressing with antioxidant properties for wound healing. Histol Histopathol. 2015 Dec;30(12):1499-512. doi: 10.14670/HH-11-646. Epub 2015 Jul 3. PMID 26140672
- [Background] Castro B, Bastida FD, Segovia T, Lopez Casanova P, Soldevilla JJ, Verdu-Soriano J. The use of an antioxidant dressing on hard-to-heal wounds: a multicentre, prospective case series. J Wound Care. 2017 Dec 2;26(12):742-750. doi: 10.12968/jowc.2017.26.12.742. PMID 29244974